CLINICAL TRIAL: NCT02723383
Title: Baclofen to Prevent Agitation in Alcohol Addicted Patients in ICU: Study Protocol for a Randomised Controlled Against Placebo Trial
Brief Title: Baclofen to Prevent Agitation in Alcohol Addicted Patients in ICU
Acronym: BACLOREA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC15_0036
Record Dates: First submitted 2016-03-03; First posted 2016-03-30 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Alcoholism
Keywords: alcoholism; intensive care; Baclofen; restlessness; Delirium tremens; Alcohol withdrawal syndrome
MeSH Terms: conditions — Alcoholism; Psychomotor Agitation; Alcohol Withdrawal Delirium | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BACLOFEN (Experimental): patient will receive baclofen caps
  Interventions: Drug: BACLOFEN
- PLACEBO (Placebo Comparator): patient will receive placebo caps (lactose)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: BACLOFEN — Daily doses will be adapted to daily MDRD creatinine clearance from 150 to 50mg. On the day of randomisation, the patient will receive the full daily dose in a one-shot administration. Then daily doses will be divided into 3 intakes on the following days. During the mechanical ventilation period, the treatment will be administered via the nasogastric feeding tube. After extubation, the treatment will be administered either via the nasogastric tube or the oral route.
  Arms: BACLOFEN
Drug: PLACEBO — Daily doses will be adapted to daily MDRD creatinine clearance from 150 to 50mg. On the day of randomisation, the patient will receive the full daily dose in a one-shot administration. Then daily doses will be divided into 3 intakes on the following days. During the mechanical ventilation period, the placebo will be administered via the nasogastric feeding tube. After extubation, the placebo will be administered either via the nasogastric tube or the oral route.
  Arms: PLACEBO

SUMMARY:
Background: Alcohol is the leading psychoactive substance consumed in France, with about 15 million regular consumers. The National institute on Alcohol Abuse and Alcoholism (NIAAA) considers alcohol abuse to be more than 14 units of alcohol a week for men and 7 units for women. The specific complication of alcoholism is the alcohol withdrawal syndrome. Its incidence reaches up to 30% and its main complications are Delirium Tremens, restlessness, extended hospital stay, higher morbidity, psychiatric and cognitive impairment. Without appropriate treatment, Delirium Tremens can lead to death in up to 50% of patients.

Methods/Design: This prospective, randomised, controlled study versus placebo will be conducted in eighteen French intensive care units (ICU). Patients with an alcohol intake higher than the NIAAA threshold, under mechanical ventilation, will be included. The primary objective is to determine whether Baclofen is more efficient than placebo in preventing restlessness-related side effects in ICU. Secondary outcomes include mechanical ventilation duration, length of ICU stay, cumulative doses of sedatives and painkillers received within 28 days of ICU admission. Restlessness-related side effects are defined as unplanned extubation, Medical disposal removal, falling out of bed, ICU runaway, immobilisation device removal, self-aggression or towards medical staff. Daily doses of Baclofen/placebo will be guided by creatinine clearance assessment once a day.

Discussion: Restlessness in alcoholic patients is a life-threatening issue in ICUs. BACLOREA is a randomised study assessing the capacity of Baclofen to prevent agitation in mechanically-ventilated patients. Enrolment of 314 patients will begin in June 2016 and is expected to end in December 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 80 years old with an estimated alcohol intake of:

  * 14 units of alcohol per week during the month before hospitalisation for men aged 18 to 64
  * 7 units of alcohol per week during the month before hospitalisation for women or men older than 65.

AND Intubated, ventilated with an expected duration of mechanical ventilation> 24 hours at least

Exclusion Criteria:

* Hospitalization > 7 days
* Baclofen administration before ICU admission (personal treatment or single administration)
* Pregnancy
* Porphyria
* Burned on ICU admission
* Personal treatment including Gamma-hydroxybutyric acid (Alcover/Xyrem)
* Recent stroke or subarachnoid haemorrhage or head trauma with radiological evidence
* Recent or old paraplegia or tetraplegia
* Cardiac arrest with resuscitation manoeuvres before or after ICU admission
* Contraindication to Enteral drug administration for longer than 24 hours
* Lack of social protection
* Hypersensitivity to Baclofen
* Coeliac disease
* Refractory epilepsy
* Dementia, schizophrenia, Bipolar disorder or severe depression.
* Parkinson's disease
* Health care limitation owing to pejorative prognosis
* Tracheotomy on ICU admission
* Patients under guardianship or trusteeship
* Patients already enrolled in interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Occurrence (yes or no) of agitation-related adverse events | at the end of treatment (22 days max)
  Occurrence (yes or no) of agitation-related adverse events during treatment/placebo administration with at least one sign out of the following:
  * Unplanned extubation
  * Medical disposal removal
  * Falling out of bed
  * ICU runaway
  * Immobilization device removal
  * Self-aggression or aggression towards medical staff.

SECONDARY OUTCOMES:
Adverse event (yes or no) related to agitation | within 28 days of ICU admission
Extubation failure defined as reintubation | within the next 48 hours after extubation
Tracheotomy for failure of mechanical ventilation weaning during hospitalization | an average of 28 days
Infections acquired in the ICU: Urinary infection, pneumonia, catheter infection or bacteraemia during hospitalization | an average of 28 days
Total doses of sedatives and painkillers received in the ICU | within 28 days of ICU admission
Riker Sedation -Agitation Scale (SAS) in the ICU | within 28 days of ICU admission
Daily CIWA-Ar alcohol withdrawal score | during the week following extubation
Duration of mechanical ventilation during hospitalization | an average of 28 days
Ventilation free days (VFD) | at day 28
Length of ICU stay | within 90 days
Length of total hospitalisation | within 90 days
Death in ICU | at days 28 and 90
Death during hospital stay during hospitalization | within 90 days
Number of adverse event (s) per patient occurring in ICU from Day 1 to Day 28 | until Day 28
Agitation requiring rapid intravenous or intramuscular administration of an hypnotic or neuroleptic (bolus) | until Day 28
Reintubation due to restlessness or withdrawal syndrome | until Day 28
Agitation and mortality in ICU at Day 28 | at Day 28

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU ANGERS - réanimation chirurgicale, Angers
  - CHU de Brest Réanimation Chirurgicale, Brest
  - CHU de Brest Réanimation Médicale, Brest
  - CHU de Caen Réanimation Médicale, Caen
  - CHD La Roche Sur YON, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - Centre Hospitalier de Bretagne Sud Réanimation Polyvalente Lorient, Lorient
  - CHU MONTPELLIER - Lapeyronie, Montpellier
  - Chu Montpellier, Montpellier
  - CHU NANTES - réanimation chirurgicale, Nantes
  - CHU NANTES -réanimation médicale, Nantes
  - Hopital Saint Antoine, Paris
  - Chu Poitiers, Poitiers
  - Ch Cornouaille, Quimper
  - Chu Rennes, Rennes
  - CHR Saint Nazaire, Saint-Nazaire
  - CHRU Tours Bretonneau, Tours
  - Chu Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vourc'h M, Garret C, Gacouin A, Lacherade JC, Jonas M, Klouche K, Ferrandiere M, Jaber S, Flet L, Dailly E, Pouplet C, Maamar A, Reignier J, Roquilly A, Feuillet F, Mahe PJ, Asehnoune K; BACLOREA study group. Effect of High-Dose Baclofen on Agitation-Related Events Among Patients With Unhealthy Alcohol Use Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2021 Feb 23;325(8):732-741. doi: 10.1001/jama.2021.0658. PMID 33620407
- [Derived] Vourc'h M, Feuillet F, Mahe PJ, Sebille V, Asehnoune K; BACLOREA trial group. Baclofen to prevent agitation in alcohol-addicted patients in the ICU: study protocol for a randomised controlled trial. Trials. 2016 Aug 19;17(1):415. doi: 10.1186/s13063-016-1539-2. PMID 27542731